CLINICAL TRIAL: NCT03417570
Title: Cap Assisted Upper Endoscopy Versus High Definition White Light Endoscopy and Narrow Band Imaging Alone In The Detection Of Visible Lesions Barrett's Esophagus: A Randomized Tandem Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 201708210
Record Dates: First submitted 2018-01-25; First posted 2018-01-31 (Actual); Results first posted 2022-07-29 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Endoscopy, Digestive System; Narrow Band Imaging; Contraceptive Devices, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm 1: EGD with cap first, followed by EGD without cap (Experimental): -Participants in the first arm will undergo EGD with cap first, followed by EGD without cap in the same procedural period.
  Interventions: Procedure: Esophagogastroduodenoscopy with high definition-white light end endoscopy (HD-WLE) and narrow band imaging (NBI); Device: Olympus Disposable Distal Attachment Cap
- Arm 2: EGD without cap first, followed by EGD with cap (Experimental): -Participants in the second arm will undergo EGD without cap first, followed by EGD with cap in the same procedural period.
  Interventions: Procedure: Esophagogastroduodenoscopy with high definition-white light end endoscopy (HD-WLE) and narrow band imaging (NBI); Device: Olympus Disposable Distal Attachment Cap

INTERVENTIONS:
Procedure: Esophagogastroduodenoscopy with high definition-white light end endoscopy (HD-WLE) and narrow band imaging (NBI) — -The second endoscopist will be blinded to the results of the initial exam.
  Other Names: EGD
Device: Olympus Disposable Distal Attachment Cap — -The second endoscopist will be blinded to the results of the initial exam.
  Other Names: Cap

SUMMARY:
The hypothesis is that the addition of a transparent cap to the end of the endoscope will increase the detection and diagnostic yield of visible lesions in Barrett's esophagus. Thus, the goal of this tandem design trial is to compare the diagnostic yield (DY) of cap assisted endoscopy with that of conventional endoscopy using high definition-white light endoscopy (HD-WLE) and narrow band imaging (NBI) in patients with Barrett's esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age.
* Must be patients undergoing standard of care EGD for the confirmation of dysplasia in BE or EET for dysplasia in BE.
* Must be able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Prior endoscopic treatment for BE.
* Unable to tolerate sedation due to medical comorbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir M Kushnir, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: EGD With Cap First, Followed by EGD Without Cap | Arm 2: EGD Without Cap First, Followed by EGD With Cap
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: EGD With Cap First, Followed by EGD Without Cap | Arm 2: EGD Without Cap First, Followed by EGD With Cap | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Full Range); unit: years] | 65.5 [30 to 85] | 66 [43 to 91] | 66 [30 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 43 | 42 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 50 | 49 | 99
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 49 | 50 | 99
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had a Diagnostic Yield Obtained
Description: -Diagnostic yield is defined as Barrett's esophagus lesions that were identified and confirmed histologically as low grade dysplasia, high grade dysplasia, intramucosal cancer, or invasive adenocarcinoma
Time Frame: At the time of procedure (day 1)
Population: Participants had to have visible lesions to be evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- EGD Without CAP: -Esophagogastroduodenoscopy (EGD) with high-definition-white light endoscopy (HD-WLE) and narrow band imaging (NBI)
- EGD With CAP: -Cap-assisted esophagogastroduodenoscopy (EGD) with high-definition-white light endoscopy (HD-WLE) and narrow band imaging (NBI)
Arm/Group | EGD Without CAP | EGD With CAP
Number analyzed (Participants) | 56 | 60
Participants | 56 | 60

2. Secondary Outcome: Number of Participants With Visible Lesions in EGD With Cap Versus Without Cap
Time Frame: At the time of procedure (day 1)
Measure: Count of Participants; unit: Participants
Arm/Group | EGD Without CAP | EGD With CAP
Number analyzed (Participants) | 100 | 100
Participants | 56 | 60

3. Secondary Outcome: Number of Participants With High Grade Dysplasia or Esophageal Adenocarcinoma
Time Frame: At the time of procedure (day 1)
Population: Out of the 100 enrolled participants, there were 2 participants with missing pathology reports.
Measure: Count of Participants; unit: Participants
Arm/Group | EGD Without CAP | EGD With CAP
Number analyzed (Participants) | 98 | 98
Participants | 22 | 23

4. Secondary Outcome: Total Procedure Duration in Seconds
Time Frame: At the time of procedure (day 1)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | EGD Without CAP | EGD With CAP
Number analyzed (Participants) | 100 | 100
seconds | 160.9 (74.6) | 159.8 (73.4)

5. Secondary Outcome: Safety as Measured by Number of Participants With Procedure-related Adverse Events
Description: * The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
  * Adverse events were collected for the entire procedure as a whole and for 48 hours after the procedure and were not separately collected for each part of the procedure (EGD without CAP versus EGD with CAP).
Time Frame: Through 48 hours after EGD
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: EGD With Cap First, Followed by EGD Without Cap | Arm 2: EGD Without Cap First, Followed by EGD With Cap
Number analyzed (Participants) | 50 | 50
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of EGD until 48 hours after EGD.
Description: Adverse events were collected for the entire procedure as a whole and for 48 hours after the procedure and were not separately collected for each part of the procedure (EGD without CAP versus EGD with CAP).
Arm/Group | Arm 1: EGD With Cap First, Followed by EGD Without Cap | Arm 2: EGD Without Cap First, Followed by EGD With Cap
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT03417570/Prot_SAP_000.pdf